CLINICAL TRIAL: NCT05580419
Title: Impact of a Novel Community-Based Biobehavioral Chronic Pain Team Training Program (4PCP) on Practitioner and Patient Outcomes
Brief Title: Impact of 4PCP on Practitioner and Patient Outcomes
Acronym: 4PCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Medical College of Wisconsin (Other); Case Western Reserve University (Other); SSM Health (Other); Wisconsin Research and Education Network (Network); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM20025110; R01HS028630 (AHRQ)
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single-blinded, stepped cluster design trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4PCP Course (for practitioners only) (Experimental): All enrolled practitioners will be assigned to take the 4PCP course as the intervention. Patients will not be assigned to the course and will only be completing surveys before and after their practitioner completes 4PCP.
  Interventions: Behavioral: 4PCP Course

INTERVENTIONS:
Behavioral: 4PCP Course — 4PCP is a training framework for the management of chronic pain and gives practitioners lasting knowledge on how to better care for chronic pain patients.

SUMMARY:
Reducing opioid prescribing and improving outcomes in patients with chronic pain would benefit our nation. Neither addiction nor chronic pain spares any race, gender, or particular socio-economic status. This study is investigating a potentially inexpensive way of providing a previously costly service (the intensive chronic pain rehabilitation program), which is why insurers stopped covering it. Although it is unusual for an application from an academic institution to include a startup company (PainSTakers, LLC) as the curriculum provider, this is actually a long-term strength of this program, and the reason NIH recommended this route. It ensures that 4PCP will ultimately sustain itself rather than require government support for its continuation. Support for this application is not to provide the curriculum, but to determine if it is effective in the outcomes expected to be found. The curriculum is being provided freely only as an incentive for practitioners to participate in the research portion of the study. If the study is able to demonstrate its clinical effectiveness, the next step will be to show a positive economic impact for health care institutions and for health insurers who may then wish to support the program for their practitioners and their patients.

DETAILED DESCRIPTION:
Practitioner procedures:

After the completion of informed consent, practitioners will be sent their first set of surveys (Baseline).

1 week before the first day of the practitioner's course, they will be sent a second set of surveys (Time 0).

6 months after course completion, practitioners will be sent their next set of surveys (Follow Up 1).

6 months after the distribution of Follow Up Survey 1, practitioners will be sent their next set of surveys (Follow Up 2).

6 months after the distribution of Follow Up Survey 2, practitioners will be sent their next set of surveys (Follow Up 3).

6 months after the distribution of Follow Up Survey 3, practitioners will be sent their final set of surveys (Follow Up 4).

Patient procedures:

After the completion of informed consent, patients will be sent their first set of surveys (Baseline).

1 week before the first day of the patient's practitioner's course, they will be sent a second set of surveys (Time 0).

6 months after their practitioner's course completion, patients will be sent their next set of surveys (Follow Up 1).

6 months after the distribution of Follow Up Survey 1, patients will be sent their next set of surveys (Follow Up 2).

6 months after the distribution of Follow Up Survey 2, patients will be sent their next set of surveys (Follow Up 3).

6 months after the distribution of Follow Up Survey 3, patients will be sent their final set of surveys (Follow Up 4).

Practitioner measures:

* Demographics
* HC-PAIRS
* Mini Z & Burnout
* PABS-PT
* Skills Comparison
* Multi-Disc Perspective Questionnaire
* CPPP (for MDs/DOs)
* Know Pain-12

Patient measures:

* Demographics
* Medication information
* PEG-3
* PCS
* PROMIS 8A
* PROMIS Global Health
* PROMIS Pain Interference
* GAD-7
* PHQ-8
* Secondary measures abstracted from state prescribing records

Practitioner interventions:

4PCP training course

Patient interventions:

No direct interventions, but concepts practitioners learn from the 4PCP curriculum may change the way the practitioner continues care with the patient.

ELIGIBILITY:
Practitioner Inclusion:

* General practitioners
* Part of a practice that has their own identifiable patient population including patients with chronic pain
* Able to fully answer questionnaires
* Able to attend 4PCP course
* English speaking

Patient inclusion:

* Age 14-80
* Self-report of chronic non-malignant pain > 3 months
* No foreseeable or planned surgeries for chronic pain
* Has attended at least 2 established visits in the enrolled practitioner's practice
* English speaking

Practitioner exclusion:

* Pain specialists
* Unable to fully answer questionnaires
* Unable to attend the 4PCP course
* Non-English speaking

Patient exclusion:

* Unable to answer questionnaires (e.g. stroke, dementia, developmental delay, etc.)
* Followed in a specialty pain clinic (PCP not managing pain care)
* Sickle cell disease
* Prisoners
* Non-English speaking

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1188 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Participant Pain, Enjoyment of Life and General Activity (PEG-3) | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  Pain, Enjoyment of Life and General Activity will be assessed using the PEG-3 which is a self-report, 3 item survey which asks patient participants to rate their experiences on a 10 point Likert scale.
Change in Practitioner Chronic Pain Physician Perspectives Questionnaire (CPPP) | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  Practitioner chronic pain perspectives will be assessed using the CPPP, which is a self-report 26 item survey that asks practitioners to rate feelings related chronic pain on a 6 point Likert scale.
Number of Patient Participants whose opioid dose tapered | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  Opioid Morphine milligram equivalents (MME) MME will be calculated from medical record/state prescription monitoring data to determine changes in patient opioid use. Based on MME changes, number of patients whose dose is tapered by at least 5% over 6 months will be counted.

SECONDARY OUTCOMES:
Change in Patient Participant Pain Catastrophizing Scale (PCS) | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  Pain catastrophization will be assessed using the PCS which is a self-report, 13 item survey which asks participants to rate how often they have the thoughts and feelings described in each item when they are in pain on a 5 point Likert scale.
Change in Patient Participant Pain Interference (PI) | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  PI will be assessed using the PROMIS Pain Interference - Short Form 8a which is a self-report, 8 item survey which asks participants to rate the degree to which pain interfered in their lives on a 5-point Likert scale.
Change in Patient Participant Quality of Life (QoL) | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  QoL will be assessed using the PROMIS Global Health Scale which is a self-report, 10 item survey which asks participants to rate their perception of their physical and mental health on a 5-point Likert Scale.
Change in Patient Participant Generalized Anxiety Disorder (GAD-7) | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  Anxiety levels will be assessed using the GAD-7 which is a self-report, 8 item survey which asks participants to rate how often they have the thoughts/feelings/behaviors described in each item on a 4 point Likert scale.
Change in Patient Participant Patient Health Questionnaire (PHQ-9) | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  Patient Health will be assessed using the PHQ-9 which is a self-report, 10 item survey which asks participants to rate how bothered they have been by physical/mental symptoms on a 4-point Likert Scale.
Change in Practitioner Health Care Providers' Pain and Impairment Relationship Scale (HC-PAIRS) | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  Practitioner pain and impairment relationship will be assessed using HC-PAIRS, which is a self-report 15 item survey that asks practitioners to answer questions about their perception on the abilities of chronic pain patients on a 7 point Likert scale.
Change in Practitioner Chronic Pain Attitudes and Beliefs Questionnaire (PABS-PT) | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  Practitioner career perspectives of chronic pain knowledge will be measured with the PABS-PT, which is a self-report 14 item survey that asks practitioners to rate their attitudes and beliefs on chronic pain care on a 6 point Likert scale.
Change in Practitioner Burn-Out (Mini Z) | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  Practitioner career burn-out perception will be assessed using the Mini Z scale, which is a self-report 10 item survey that asks practitioners to rate feelings related to burn-out on a 5 point Likert scale. This measure differs from the Burn-Out measure in Outcome 7 because it includes the addition of questions relating to workplace environment.
Practitioner Burn-Out | Upon enrollment, 1 week before practitioner course participation, up to 3 years after practitioner course participation
  Practitioner career burn-out perception will be assessed using the Practitioner Burn-Out scale, which is a self-report 3 item survey that asks practitioners to rate feelings related to burn-out on a 10 point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chelimsky, M.D., Principal Investigator — VCU
Locations (4):
- United States (4):
  - Case Western Reserve University, Cleveland, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
  - Wisconsin Research and Education Network (WREN), Madison, Wisconsin
  - SSM Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Only de-identified aggregate data will be shared with other researchers.

REFERENCES:
- [Background] Chelimsky TC, Fischer RL, Levin JB, Cheren MI, Marsh SK, Janata JW. The primary practice physician program for chronic pain ((c) 4PCP): outcomes of a primary physician-pain specialist collaboration for community-based training and support. Clin J Pain. 2013 Dec;29(12):1036-43. doi: 10.1097/AJP.0b013e3182851584. PMID 23459398
- [Background] Why the US Should Develop a Primary Medical Specialty in Pain Medicine. American Board of Pain Medicine [Web]; Available from: http://abpm.org/uploads/files/talking%20points%20-%20federal%20approach%20needed%20final.pdf
- [Background] Okumura MJ, Heisler M, Davis MM, Cabana MD, Demonner S, Kerr EA. Comfort of general internists and general pediatricians in providing care for young adults with chronic illnesses of childhood. J Gen Intern Med. 2008 Oct;23(10):1621-7. doi: 10.1007/s11606-008-0716-8. Epub 2008 Jul 26. PMID 18661191
- [Background] Aydede M, Shriver A. Recently introduced definition of "nociplastic pain" by the International Association for the Study of Pain needs better formulation. Pain. 2018 Jun;159(6):1176-1177. doi: 10.1097/j.pain.0000000000001184. No abstract available. PMID 29768305